CLINICAL TRIAL: NCT05628142
Title: Prospective, Multi-Center, Single Arm Post-Market Study of the Tenon Medical CATAMARAN™ SI Joint Fusion System.
Brief Title: Tenon Medical CATAMARAN™ SI Joint Fusion System CT Scan Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tenon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTL016
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Sacroiliac Joint Disruption; Degenerative Sacroiliitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CATAMARAN SI Joint Fusion System (Other): Subjects previously treated with the CATAMARAN Fixation Device
  Interventions: Radiation: Pelvic CT Scan

INTERVENTIONS:
Radiation: Pelvic CT Scan — Pelvic CT-Scan between 6-12 months post-op

SUMMARY:
The objective of this study is to evaluate 6-to-12-month radiographic outcomes of patients with sacroiliac joint disruptions or degenerative sacroiliitis that have already undergone treatment with the CATAMARAN SI Joint Fusion System. In addition, retrospective and prospective clinical outcomes will be evaluated.

DETAILED DESCRIPTION:
Patients with degenerative sacroiliitis or sacroiliac joint disruption who already had the CATAMARAN Fixation Device implanted between 6 and 12 months will be asked to return for follow-up visit to evaluate clinical outcomes and undergo a high resolution pelvic CT-Scan to assess fusion. Additionally, retrospective clinical outcomes will be collected from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years of age at time of treatment with the CATAMARAN SI Joint Fusion System
* Patient implanted with the CATAMARAN Fixation Device within the last 12 months
* Diagnosis of sacroiliac joint disruption or degenerative sacroiliitis
* Patient, or authorized representative, signs a written Informed Consent form to participate in the study
* Patient is willing and able to complete study follow-up requirements

Exclusion Criteria:

* Known or suspected active drug or alcohol abuse
* Previously diagnosed osteoporosis (defined as prior T-score <-2.5 or history of osteoporotic fracture) or prior/current use of drug therapy for osteoporosis.
* Prior fracture of any bone related to cancer/tumor (i.e., pathologic fracture)
* Prior diagnosis of tumor in sacrum or ilium
* Unstable fracture of sacrum and or ilium involving the targeted SIJ
* Osteomalacia or other metabolic bone disease
* Use of medications known to have detrimental effects on bone quality and soft-tissue healing
* Patient is pregnant or wishes to become pregnant during the study period
* Patient is not likely to comply with the follow-up evaluation schedule
* Patient is a prisoner or a ward of the state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Radiographic Fusion | 6-12 month post CATAMARAN Fixation Device implantation
  The primary endpoint is the proportion of subjects that demonstrate radiographic fusion assessed by CT-Scan, as evaluated by an Independent Radiologist.

SECONDARY OUTCOMES:
Device Status | 6-12 months post-op
  Radiographic assessment for device status: device placement, loosening, migration and/or breakage
Surgical re-intervention for SI joint pain | 6-12 months post-op
  Proportion of patients requiring surgical re-intervention (removal, revision, reoperation, or supplemental fixation) for SI joint pain
Neurologic worsening related to the sacral spine | 6-12 months post-op
  Proportion of patients experiencing neurologic worsening related to the sacral spine compared to baseline
Serious device related adverse events | 6-12 months post-op
  Summary of all serious device related adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Minimally Invasive Neurosurgery of Texas, Plano, Texas
  - St. George Orthopaedic Spine, St. George, Utah

IPD SHARING:
Plan to Share IPD: No